CLINICAL TRIAL: NCT01841593
Title: A Two Way Cross Over Pharmacokinetic (PK) Interaction Study Between Raltegravir and Amlodipine in Healthy Volunteers
Brief Title: A Two Way Cross Over Pharmacokinetic Interaction Study Between Raltegravir and Amlodipine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SSAT 051
Record Dates: First submitted 2013-04-16; First posted 2013-04-26 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: HIV
MeSH Terms: interventions — Raltegravir Potassium; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): DAYS 1 to 7: raltegravir 400 mg BID DAYS 8 to 14: raltegravir 400 mg BID PLUS amlodipine 5 mg OD DAYS 15 to 21: amlodipine 5 mg OD
  Interventions: Drug: Raltegravir; Drug: Amlodipine
- Group B (Experimental): DAYS 1 to 7: amlodipine 5 mg OD DAYS 8 to 14: raltegravir 400 mg BID PLUS amlodipine 5 mg OD DAYS 15 to 21: raltegravir 400 mg BID
  Interventions: Drug: Raltegravir; Drug: Amlodipine

INTERVENTIONS:
Drug: Raltegravir — Isentress 400mg tablet taken twice daily
  Other Names: Isentress
Drug: Amlodipine — generic amlodipine 5mg tablets (Accord healthcare Limited, UK)
  Other Names: Amlodipine 5mg tablets

SUMMARY:
The purpose of the study is to look at the levels of an HIV medication (raltegravir) in the blood, and how it is affected if raltegravir is taken at the same time as another medicine for high blood pressure (amlodipine). Many patients with HIV will also have high blood pressure, so it is important to know which drugs for each of these conditions can be taken together without affecting how well they work individually.

Over a 3 week period, participants took amlodipine for 2 weeks, and raltegravir for 2 weeks, with the middle week being on both drugs. The investigators will look at and compare the levels of these two drugs in the blood after subjects have taken them separately and both together.

This study is randomised into two groups with both study medications received by all participants in a three-period crossover pattern; randomisation determined which medication was taken first. Once randomised allocation was performed, medications were administered in an open-label fashion.

DETAILED DESCRIPTION:
HIV-negative male and female volunteers will be enrolled, after written confirmation of informed consent, in a phase I, open-label, cross-over, PK study (approved by Westminster Research Ethics Committee and UK Regulatory Authorities; Eudra number 2012-005400-18).

Subjects are randomized to receive either raltegravir 400mg twice-daily (seven days), followed by raltegravir 400mg twice-daily plus amlodipine 5mg once-daily (seven days), followed by amlodipine 5mg once-daily alone (seven days), or the same treatments in the opposite order, in the fasted state (at least eight hours) with 240mL of water.

Intensive PK sampling and safety laboratory analysis are performed at the end of each phase (Days 7, 14 and 21). Raltegravir and amlodipine plasma concentrations will be analysed by a validated liquid chromatography-mass spectrometry (LC-MS/MS) method.

PK parameters are determined by non-compartmental methods [WinNonlin Phoenix (version 6.1; Pharsight Corp, Mountain View, CA, USA]. These are the concentrations measured 12 and 24 hours post-dose (C12h, C24h) for raltegravir and amlodipine, respectively; the maximum concentration (Cmax); and the area under the curve over 12 and 24 hours (AUC12h, AUC24h) for raltegravir and amlodipine, respectively.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria within 28 days prior to the baseline visit:

* The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements
* Male or non-pregnant, non-lactating females
* Between 18 to 65 years, inclusive
* Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 12 weeks after the study
* Willing to consent to their personal details being entered onto The Over-volunteering Prevention Scheme (TOPS) database
* Willing to provide photographic identification at each visit.
* Registered with a GP in the UK

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

* Any significant acute or chronic medical illness including hypertension (BP persistently >140/90 mmHg) or hypotension (BP persistently <90/60 mmHg)
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
* Positive blood screen for hepatitis B surface antigen and/or C antibodies
* Positive blood screen for HIV-1 and/or 2 antibodies
* Current or recent (within 3 months) gastrointestinal disease
* Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study
* Exposure to any investigational drug or placebo within 3 months of first dose of study drug
* Use of any other drugs (unless approved by the Investigator), including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug, unless approved/prescribed by the Principal Investigator as known not to interact with study drugs.
* Females of childbearing potential without the use of effective non-hormonal birth control methods, or not willing to continue practising these birth control methods for at least 12 weeks after the end of the treatment period
* Previous allergy to any of the constituents of the pharmaceuticals administered in this trial
* Lactose intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's AIDS Trust, London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (Raltegravir Then Amlodipine): DAYS 1 to 7: raltegravir 400 mg BID DAYS 8 to 14: raltegravir 400 mg BID PLUS amlodipine 5 mg OD DAYS 15 to 21: amlodipine 5 mg OD
- Group B (Amlodipine Then Raltegravir): DAYS 1 to 7: amlodipine 5 mg OD DAYS 8 to 14: raltegravir 400 mg BID PLUS amlodipine 5 mg OD DAYS 15 to 21: raltegravir 400 mg BID
Period: First Intervention (Days 1 to 7)
Arm/Group | Group A (Raltegravir Then Amlodipine) | Group B (Amlodipine Then Raltegravir)
Started | 12 | 7
Completed | 12 | 6
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Second Intervention (Days 8 to 14)
Arm/Group | Group A (Raltegravir Then Amlodipine) | Group B (Amlodipine Then Raltegravir)
Started | 12 | 6
Completed | 11 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Third Intervention (Days 15 to 21)
Arm/Group | Group A (Raltegravir Then Amlodipine) | Group B (Amlodipine Then Raltegravir)
Started | 11 | 6
Completed | 11 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who completed at least two of three pharmacokinetic sessions for comparison were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 6 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Raltegravir and Amlodipine Without and With Co-administration of the Other Studied Drug.
Description: To investigate the pharmacokinetics of raltegravir and amlodipine co-administration. The pharmacokinetic parameters calculated for raltegravir and amlodipine will be trough concentration (Ctrough), defined as the concentration at 24 hours after the observed drug dose, the maximum observed plasma concentration (Cmax), elimination half-life (t1/2), time point at Cmax (Tmax), and total drug exposure, expressed as the area under the plasma concentration-time curve from 0-24 hours after dosing (AUC0-24h).
  All pharmacokinetic parameters will be calculated using non-compartmental modeling techniques (WinNonlin®) and all statistical calculations performed and analyzed using SAS version 9.1 or SPSS V17.0.
Time Frame: Day 7 of each intervention (0 (pre-dose), 2, 4, 8 and 12 hours post dose (both drugs) and 24 hours post dose (amlodipine only))
Population: Data from all enrolled participants who participated in at least two of the three PK assessments were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Raltegravir PK (Alone); Raltegravir PK (Administered With Amlodipine); Amlodipine PK (Alone); Amlodipine PK (Administered With Raltegravir): Combined analysis - groups A & B. No period effect due to order of study treatment periods found.
Arm/Group | Raltegravir PK (Alone) | Raltegravir PK (Administered With Amlodipine) | Amlodipine PK (Alone) | Amlodipine PK (Administered With Raltegravir)
Number analyzed (Participants) | 17 | 17 | 17 | 17
ng/mL | 1178 [966 to 2318] | 1866 [1779 to 4511] | 8.47 [7.58 to 10.0] | 8.49 [7.65 to 9.94]

2. Primary Outcome: Raltegravir C12h
Description: measured concentration 12 hours after dose in the absence, and presence, of amlodipine.
Time Frame: 12 hours post-dose on day 7 of daily dosing.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Raltegravir PK (Alone) | Raltegravir PK (Administered With Amlodipine)
Number analyzed (Participants) | 17 | 17
ng/mL | 48 [35 to 95] | 37 [30 to 67]

3. Primary Outcome: Amlodipine C24h
Description: measured concentration 24 hours after dose in the absence, and presence, of raltegravir
Time Frame: 12 hours post-dose on day 7 of daily dosing.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Amlodipine PK (Alone) | Amlodipine PK (Administered With Raltegravir)
Number analyzed (Participants) | 17 | 17
ng/mL | 4.91 [4.23 to 6.36] | 4.55 [4.11 to 5.34]

4. Primary Outcome: Raltegravir AUC(0-12h )
Description: AUC0-12h: Area under the concentration time curve over 12 hours in the absence, and presence, of amlodipine.
Time Frame: Post dose after day 7 of daily dosing
Measure: Geometric Mean (95% Confidence Interval); unit: ng*h/mL
Arm/Group | Raltegravir PK (Alone) | Raltegravir PK (Administered With Amlodipine)
Number analyzed (Participants) | 17 | 17
ng*h/mL | 4600 [3888 to 7652] | 6410 [5649 to 12138]

5. Primary Outcome: Amlodipine AUC(0-24h)
Description: AUC0-24h: Area under the concentration time curve 24 hours in the absence, and presence, of raltegravir
Time Frame: Post-dose on day 7 of daily dosing
Measure: Geometric Mean (95% Confidence Interval); unit: ng*h/mL
Arm/Group | Amlodipine PK (Alone) | Amlodipine PK (Administered With Raltegravir)
Number analyzed (Participants) | 17 | 17
ng*h/mL | 166.0 [146.3 to 202.9] | 165.9 [148.7 to 195.8]

ADVERSE EVENTS:
Time Frame: Event data collected from time of signing informed consent at screen, until discharge from study (14 days after completion).
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/7
Other Adverse Events (participants affected / at risk) | 6/12 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=12) | Group B (N=7)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=12) | Group B (N=7)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
gingivitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
pruritic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
pedal oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
insect bite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
light-headed (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes